CLINICAL TRIAL: NCT05949112
Title: Efficacy of Manual or Mechanical Toothbrush in the Genesis and Prevention of Dental
Brief Title: Toothbrush in the Genesis and Prevention of Dental Recessions
Acronym: Recession
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Paolo Pesce, Prof, Universita degli Studi di Genova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Recession1
Record Dates: First submitted 2023-06-27; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Recession, Gingival
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual (Experimental): Manual toothbrush
  Interventions: Device: soft bristle toothbrush
- Mechanical (Experimental): Mechanical toothbrush
  Interventions: Device: mechanical toothbrush

INTERVENTIONS:
Device: soft bristle toothbrush — manual toothbrushes
  Arms: Manual
Device: mechanical toothbrush — sonic toothbrush
  Arms: Mechanical

SUMMARY:
The aim of this research is to evaluate the effect of brushing on gingival recessions and to understand the impact of manual brushing and brushing with mechanical aid on their evolution.

The study involves the recruitment of 90 patients with or without gingival recessions at the Dentistry service of the University of Genoa.

The first phase involves the evaluation of the brushing force on the genesis of gingival recessions. A questionnaire will be filled out and the same toothbrushes and toothpastes will be provided for one month to 30 patients with recessions and 30 patients without recessions. After a month, the "wear" of the manual toothbrush and the gingival health indices will be measured.

In this phase 60 patients with recessions will be divided into two groups according to the oral hygiene method that will be recommended. In the first group a super soft toothbrush will be delivered, in the second group a mechanical toothbrush. Gingival health indices will be taken and an intraoral scan will be done to measure recessions. At 6 months and 12 months the indices will be measured again and compared between the two groups.

This research has two objectives:

1. Evaluate the differences in wear of the manual toothbrush head after one month of use between patients with gum recession and patients without gum recession. In the case of greater wear among patients with recessions it could be assumed that a greater brushing force is able to determine the formation of recessions.
2. Try to understand if there are differences between the super soft manual toothbrush and the mechanical toothbrush regarding the effectiveness of use and the "delicacy" on recession. Both tools are currently recommended for patients with recessions, but there are no studies in the literature comparing the two tools.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old;
* Fully dentate participants;
* Periodontal health

Exclusion Criteria:

* Patient with periodontitis
* Previous ortho treatment
* Insufficient restorations or prostheses.
* Systemic disease affecting the periodontal tissues (e.g. bleeding disorders, diabetes mellitus etc.)
* Patients under medication associated with gingival enlargement (e.g. calcium channel blockers, immunosuppressants or anticonvulsants).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-27 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change of Gengival recession from baseline to 6 months | 0-6 months
  gingival recession
Change of Gengival recession from baseline to 12 months | 0-12 months
  gingival recession

SECONDARY OUTCOMES:
FMPS | 6 months
  full moth plaque score measured on 6 surfaces each tooth - percentage value
FMPS | 12 months
  full moth plaque score measured on 6 surfaces each tooth - percentage value
FMBS | 6 months
  full moth bleeding score measured on 6 surfaces each tooth - percentage value
FMBS | 12 months
  full moth bleeding score measured on 6 surfaces each tooth - percentage value

CONTACTS AND LOCATIONS:
Locations (1):
- PAD 4 ospedale san martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Undecided